CLINICAL TRIAL: NCT04655495
Title: Impact of a Low-FODMAP Gluten-free Diet on Gut Microbiota and Circulating miRNAs in Different Phenotypes of Celiac Disease Patients
Brief Title: Impact of a Low-FODMAP Gluten-free Diet on Gut Microbiota and Circulating miRNAs in Celiac Disease Patients
Acronym: FODMAP2019
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: parere 89_2019
Record Dates: First submitted 2020-11-17; First posted 2020-12-07 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Celiac Disease
Keywords: FODMAPs diet; celiac disease; microbiota; miRNA
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low FODMAPs /balanced gluten free diet (Experimental): Dietary Supplement: Balanced low FODMAPs /gluten free diet. An expert in nutrition will give a balanced gluten free diet to patients, low in FODMAPs foods.
  Interventions: Dietary Supplement: Low FODMAPs /balanced gluten free diet
- Balanced gluten free diet (Active Comparator): Balanced gluten free diet. An expert in nutrition will give a balanced gluten free diet to patients.
  Interventions: Dietary Supplement: Low FODMAPs /balanced gluten free diet

INTERVENTIONS:
Dietary Supplement: Low FODMAPs /balanced gluten free diet — Dietary Supplement: Balanced low FODMAPs /gluten free diet

SUMMARY:
15 patients with refractory celiac disease (RCD) and 15 patients with CD responsive to the GFD between the ages of 21 and 60 will be enrolled. The aim of the research will be: 1) to characterize the intestinal, blood and duodenal microbiota, then to evaluate both the taxonomy of the identified bacteria and their relative abundance 2) to analyse the profile of miRNAs from biopsy and fibroblasts isolated in the first duodenal portion, highlighting any basal deregulation and, for fibroblasts, after treatment with the 33-mer immunogenic peptide 3) quantify and know the composition of the fecal microbiota in celiac patients with persistent symptoms and in refractory celiac patients before (T0) and after (T28) treatment with a low-FODMAP diet. The aim of the study is to observe a diversification of the microbiota pattern of refractory patients vs. normoresponsive celiac patients and to observe a deregulation in the expression of miRNAs, both basally on biopsies and after treatment with the immunogenic peptide in primary fibroblast cultures.

DETAILED DESCRIPTION:
Celiac disease (CD) is a chronic, autoimmune, multisystemic disorder caused by ingestion of gluten contained in wheat. A chronic gluten-free diet (GFD) is the only therapy for CD, however a small subgroup of patients is refractory to a GFD, in fact the pathology does not regress even with a strict diet. The microbiota plays a fundamental role in the CD, in fact, especially intestinal homeostasis requires balanced interactions between the microbiota, food antigens and the host. It is widely recognized that intestinal microbiota plays a role in the initiation and progression of intestinal inflammation in numerous chronic conditions, but recent studies have shown that even the blood microbiota plays a fundamental role in autoimmune diseases. Also microRNAs (miRNAs), RNA sequences of 20-22 non-coding nucleotides that post-transcriptionally regulate gene expression, are molecules of interest in many common diseases and therefore also in CD. Fermentable, Oligo-, Di-, Mono-saccharides And Polyol (FODMAP) are short-chain carbohydrates with poor absorption in the small intestine which increases gas production and intestinal osmolarity, which can trigger gastrointestinal symptoms in sensitive individuals. A diet low in FODMAPs is a new dietary option for the treatment of persistent gastrointestinal symptoms in celiac patients. Evaluating the effect of this type of diet on intestinal microbiota changes and miRNA expression in celiac patients with persistent gastroenterological symptoms and in patients with refractory celiac disease represents an opportunity to understand how this dietary modification could contribute to the development of this disease.

15 patients with refractory celiac disease (RCD) and 15 patients with CD responsive to the GFD between the ages of 21 and 60 will be enrolled. The aim of the research will be: 1) to characterize the intestinal, blood and duodenal microbiota, then to evaluate both the taxonomy of the identified bacteria and their relative abundance 2) to analyse the profile of miRNAs from biopsy and fibroblasts isolated in the first duodenal portion, highlighting any basal deregulation and, for fibroblasts, after treatment with the 33-mer immunogenic peptide 3) quantify and know the composition of the fecal microbiota in celiac patients with persistent symptoms and in refractory celiac patients before (T0) and after (T28) treatment with a low-FODMAP diet. The aim of the study is to observe a diversification of the microbiota pattern of refractory patients vs. normoresponsive celiac patients and to observe a deregulation in the expression of miRNAs, both basally on biopsies and after treatment with the immunogenic peptide in primary fibroblast cultures.

ELIGIBILITY:
Inclusion Criteria:

* patients on a proper gluten-free diet (assessing adherence to the gluten-free diet using the Celiac Dietary Adherence Test (CDAT)
* celiac subjects diagnosed through a positive serological test of anti-endomysium antibodies (EMA) and tissue transglutaminase antibodies (TTG) evaluated through a histological abnormality in duodenal biopsies in accordance with Marsh's modified classification
* refractory celiac disease (CD)

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Subjects who follow special diets: vegetarianism, veganism
* Subjects with psychiatric disorders, diabetes mellitus, autoimmune systemic diseases, previous anaphylactic episodes, systemic disorders
* individual intolerance to disaccharides evaluated through the expired hydrogen test (lactose and fructose)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-06 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Estimated)

PRIMARY OUTCOMES:
Microbiota alpha and beta diversity | 28 days
  Evaluate both the biodiversity and the relative abundance of haematic, intestinal and duodenal bacteria in the refractory celiac population of type I and II compared to normoresponsive celiac patients

SECONDARY OUTCOMES:
miRNAs | 28 days
  Evaluate the regulation of duodenal miRNAs in RCD patients and compare them with the miRNAs expressed in normoresponsive patients
IBS symptoms | 28 days
  Improvement of VAS values of IBS symptoms in patients undergoing a balanced Gluten Free/low FODMAPs diet compared to patients undergoing only a balanced. Evaluated IBS symptoms are: abdominal pain, bloating, satisfaction with stool consistency, epigastric pain, postprandial fullness, early satiety.
SF-36 | 28 days
  Improvement of quality of life assessed through SF-36 questionnaire (eight scale scores) in patients undergoing a balanced Gluten Free/low FODMAPs diet compared to patients undergoing only a balanced gluten free diet.
SCL 90 | 28 days
  Improvement of psychological problems and symptoms of psychopathology through the symptom checklist 90 R (SCL 90 R) in patients undergoing a balanced Gluten Free/low FODMAPs diet compared to patients undergoing only a balanced gluten free diet
Dietary intake | 28 days
  Evaluation of the dietary intake in micro and macro-nutrients before and after following the assigned diet through questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Leda Roncoroni, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marasco G, Di Biase AR, Schiumerini R, Eusebi LH, Iughetti L, Ravaioli F, Scaioli E, Colecchia A, Festi D. Gut Microbiota and Celiac Disease. Dig Dis Sci. 2016 Jun;61(6):1461-72. doi: 10.1007/s10620-015-4020-2. Epub 2016 Jan 2. PMID 26725064
- [Result] Wacklin P, Laurikka P, Lindfors K, Collin P, Salmi T, Lahdeaho ML, Saavalainen P, Maki M, Matto J, Kurppa K, Kaukinen K. Altered duodenal microbiota composition in celiac disease patients suffering from persistent symptoms on a long-term gluten-free diet. Am J Gastroenterol. 2014 Dec;109(12):1933-41. doi: 10.1038/ajg.2014.355. Epub 2014 Nov 18. PMID 25403367
- See also: Results Reference — https://doi.org/10.1016/j.humic.2018.12.001